CLINICAL TRIAL: NCT03208972
Title: Prospective Randomized Trial Comparing Ovarian Stimulation in IVF-patients With Corifollitropin Alfa in Combination With Hp-FSH Versus Corifollitropin Alfa in Combination With Low Dose hCG
Brief Title: Elonva in Combination With Hp-FSH Versus Elonva With Low Dose hCG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AZ Jan Palfijn Gent (Other)
Collaborators: Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Dr. Decleer Wim, Principal Investigator, AZ Jan Palfijn Gent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-005676-34
Record Dates: First submitted 2014-05-07; First posted 2017-07-06 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Infertility
Keywords: IVF; ovarian stimulation; low dose hCG; hp-FSH; Corifollitropin Alfa; costs of IVF
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin; Menotropins; follicle stimulating hormone, human, with HCG C-terminal peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- low dose hCG (Pregnyl) (Experimental): Corifollitropin Alfa (Elonva) dosage depending on weight once administered first day of ovarian stimulation in combination 150IU low dose hCG from day 7 until final oocyte maturation.
  Interventions: Drug: low dose hCG; Drug: Corifollitropin Alfa
- hp-FSH (Menopur) (Active Comparator): Corifollitropin Alfa (Elonva) dosage depending on weight once administered first day of ovarian stimulation in combination with hp-FSH until final oocyte maturation.
  Interventions: Drug: hp-FSH; Drug: Corifollitropin Alfa

INTERVENTIONS:
Drug: low dose hCG
  Other Names: Pregnyl
  Arms: low dose hCG (Pregnyl)
Drug: hp-FSH
  Other Names: Menopur
  Arms: hp-FSH (Menopur)
Drug: Corifollitropin Alfa — Corifollitropin Alfa (Elonva) dosage depending on weight, once administered first day of ovarian stimulation for all subjects, and on day 7 they proceed with the treatment of the allocated group.
  <60 kg: Elonva 100 MCG > 60 kg: Elonva 150 MCG
  Other Names: Elonva

SUMMARY:
The study compares in a randomized controlled way two stimulation methods. One of these stimulation methods implements a new insight in ovarian follicular growth. If this novel method of stimulation proves to be as efficient as the classical stimulation protocols, there might be a dramatic reduction of the costs of the medical therapy in IVF, thus reducing also the overall IVf costs significantly.

ELIGIBILITY:
Inclusion Criteria:

* IVF/ICSI patients
* Cycle 1, 2, 3, 4

Exclusion Criteria:

* PCOS
* Endocrinological diseases

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2014-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The financial costs of the stimulation in both groups | 1 year

SECONDARY OUTCOMES:
The number of MII oocytes obtained at the occasion of the oocyte retrieval | 3 weeks
pregnancy rate | 5 weeks
duration of the stimulation | one month
hormonal levels reached at time of induction of final maturation of the oocyte | 3 weeks
the number of clinical OHSS patients | one month

CONTACTS AND LOCATIONS:
Overall Officials: Wim Decleer, MD, Principal Investigator — FERTILITY CENTER AZ JAN PALFIJN
Locations (1):
- AZ Jan Palfijn, Ghent, Oost-Vlaanderen, Belgium